CLINICAL TRIAL: NCT04878978
Title: A Randomised Study of a Personalised Approach to the Management of Preterm Rupture of Membranes and Threatened Preterm Labour
Brief Title: Premature Rupture Membranes and tPTL: a Personalised Approach (PROMPT)
Acronym: PROMPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C&W20/21
Record Dates: First submitted 2021-04-20; First posted 2021-05-10 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-04

CONDITIONS: Preterm Rupture of Membranes; Threatened Preterm Labor
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Amniocentesis

STUDY DESIGN:
Intervention Model Description: This is a single centre open labelled randomised study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (Active Comparator): Women who present with PPROM or threatened PTL and have routine care
  Interventions: Other: Routine care without amniocentesis
- Amniocentesis and biofire directed antibiotic use (Experimental): Women who present with PPROM or threatened PTL and randomised to amniocentesis and biofire directed antibiotic treatment
  Interventions: Diagnostic Test: Amniocentesis

INTERVENTIONS:
Diagnostic Test: Amniocentesis — Amniocentesis will be used to sample the amniotic fluid for Biofire detection of microorganism and to direct antibiotic treatment
  Arms: Amniocentesis and biofire directed antibiotic use
Other: Routine care without amniocentesis — Routine clinical care
  Arms: Routine care

SUMMARY:
Preterm birth (less than 37 weeks) affect approximately 8% of babies in the UK and is the worldwide leading cause of death in children under the age of 5. Subclinical infection affects approximately 50% of women giving birth before 32 weeks. Infection contributes to significant neonatal morbidity and mortality. Antibiotics such as erythromycin is currently used to treat women who present with preterm rupture of membranes. While this has shown short-term improvement in neonatal morbidity, it has not had any impact in reducing the perinatal mortality and also little effect on the health of the children at age seven. Some antibiotics such as co-amoxiclav has not shown to be effective in delaying delivery and some studies have shown that antibiotics increases rather than reduces the risk of cerebral palsy. Many women do not display signs of infection and the underlying bacteria is multifactorial (bacterial vaginosis, trichomoniasis, gonorrhoea, Chlamydia, ureaplasma, Group B streptococcal and E. Coli) and remains a diagnostic challenge. The only available clinical approach is to test the sample of amniotic fluid for bacteria and small case series have shown prolongation of pregnancy when accurately targeted antibiotic treatment is used.

This research aims to prove that targeted antibiotic therapy results in a greater prolongation of pregnancy than standard management for women with preterm prelabour rupture of membranes (PPROM) and/or threatened preterm labour (tPTL).

Women will be randomised to standard care versus BioFire directed antibiotic treatment in addition to standard care. Investigators will use the BioFire point of care testing to identify the presence of infection and identify with anti-microbial resistance genes the bacteria possess to guide the antibiotic treatment. To be certain that the presence of infection is detected the investigators will use PCR to test the amniotic fluid for IL-6 and white cell count.

DETAILED DESCRIPTION:
Overall 10-15% of women delivering before 37 weeks have intraamniotic infection and of those delivering before 32 weeks have 50% chance. Consequently, since infection is one of the most important causes of spontaneous PTL it is possible that antibiotic treatment may delay delivery and reduce the risk of fetal damage and consequently long-term disability. However, most cases do not display typical symptoms or signs of infection, the only way to make the diagnosis reliably is through performing an amniocentesis. The risk of this procedure is low in the 3rd trimester and should be considered particularly in those in PTL at less than 32 weeks, when the risk of infection is high. Studies in non-human primate models of intra-amniotic infection support for this approach, showing that specific antibiotic therapy can prevent infection-induced PTL and prolong pregnancy with improved neonatal outcomes.

Human studies have been less positive, with antibiotics failing to prolong pregnancy in PTL or eradicate infection in PPROM. The Oracle trial assessed the ability of two antibiotics, erythromycin and co-amoxiclav, to reduce the risk of PTD in women with PPROM using a composite primary outcome of neonatal death, chronic lung disease, or major cerebral abnormality on ultrasonography before discharge from hospital. Erythromycin, but not co-amoxiclav, reduced the risk of the primary outcome.

Two recent papers have challenged this negative view of the use of antibiotics for intraamniotic infection. In the first, amniocentesis was performed to identify infection or inflammation and broad-spectrum antibiotics administered to women with a singleton pregnancy presenting with tPTL at between 20 and 34 weeks. Infection was thought to be present in at least 60% of cases as judged by the presence of a raised WCC, although only 20% had positive cultures using standard microbiological approaches. 100% had an elevated IL-6 level confirming inflammation. Repeat amniocentesis confirmed resolution of inflammation in all cases and overall average prolongation was 11.4 days. In a control group not given antibiotics average prolongation was 3 days. In 3 cases infection was shown to be cleared by antibiotic treatment. In the second report, women undergoing rescue cerclage had an amniocentesis and those found to have evidence of infection or inflammation treated with broad spectrum antibiotics. A repeat amniocentesis demonstrated resolution of infection/inflammation with antibiotic treatment.

Investigators plan to recruit women to a multicenter randomised trial of standard management vs. amniocentesis with the use of BioFire filmArray point of care testing to identify the presence of bacteria and identify common anti-microbial resistance genes the bacteria possess to guide the selection of an additional antibiotic agent.

The BioFire filmArray clinical application is currently being studied in patients with pneumonia in the INHALE study. Investigators plan to use the BioFire filmArray in a maternity setting and will use the information generated by the BioFire filmArray platform to give targeted antibiotics in the amniocentesis arm in addition to routine erythromycin with the aim of prolonging latency to delivery and of improving neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 23+0 weeks and 34 weeks gestation.
2. Admitted with signs and symptoms of threatened PTL with positive fetal fibronectin of 200ng/mL or clinical confirmation of preterm rupture of membranes
3. Singleton pregnancy
4. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
5. Women must be aged 18 years or older.

   -

Exclusion Criteria:

1. Chorioamnionitis: Defined as maternal temperature was elevated to 37.8°C and two or more of the following criteria were present: uterine tenderness, malodorous vaginal discharge, maternal leucocytosis (>15 000 cells/mm3), maternal tachycardia (>100 beats/min) and fetal tachycardia (>160 beats/min).
2. Multiple pregnancy
3. Uterine contractions >2:10 and evidence on tocogram
4. Maternal infections such as HIV and hepatitis
5. Clinical suspicion of placental abruption
6. Evidence of meconium stained liquor
7. Fetal abnormality or growth restriction
8. Abnormal fetal heart rate pattern
9. Maternal pathologies in which preterm termination of pregnancy is required.

   -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The length of latency of women receiving amniocentesis with BioFire filmArray POC test guided antibiotic selection compared to those receiving standard treatment. | 4 years
  Days

SECONDARY OUTCOMES:
Maternal outcome | 4 years
  The number of women with (i) clinical diagnosis of infection including: chorioamnionitis (one or more of pyrexia, abdominal pain/tenderness, tachycardia, vaginal discharge) or (ii) postpartum endometritis with laboratory diagnosis (raised peripheral blood CRP and/or WCC, positive blood, vaginal or urine cultures)
Neonatal outcome | 4 years
  We will use a composite severe neonatal outcome of neonatal death, major adverse outcome ie, chronic lung disease (defined as the need for supplementary oxygen at 36 weeks post conception) major cerebral abnormality on ultrasonography identified prior to discharge or necrotising enterocolitis.
Microbiota and inflammatory marker endpoints | 4 years
  Maternal (vaginal, rectal, amniotic fluid) and neonatal (faecal) (measured using BioFire PCR, 16srRNA sequencing, multiplex ELISA, and associated clinical tests). Residual sample stored for future peptide/proteomics testing (e.g. MALDI-TOF multiplex). Incidence of antibiotic resistance (neonatal and maternal).
Patient based endpoints | 5 years
  Acceptability of having an amniocentesis; how risks communicated and understood; how test presented; how was the situation understood by the researchers/care givers and how did that impact on the subject's ability to understand what was being proposed? Partner perceptions and sense of inclusion/involvement.
  • Clinical data including previous obstetric history, demographic and socio-economic data and neonatal health data, the gestational age and cervical dilatation at randomisation, other drugs prescribed (corticosteroids, indomethacin, nifedipine, magnesium sulphate) will be collected.
Timing of birth | 4 years
  Number of women who deliver within 2 days
Mode of delivery | 5 years
  Vaginal, caesarean or assisted birth
Length of hospitalisation | 4 years
  Number of days of maternal hospitalisation
Gestational age at delivery | 4 years
  Weeks
Outcomes for neonates admitted to NICU | 4 years
  Number of neonates (i) admitted to NICU, (ii) ventilated, (iii) needing oxygen (iv) respiratory distress syndrome; (v) treatment with exogenous surfactant and (vi) with infection